CLINICAL TRIAL: NCT00330174
Title: The Use of Acamprosate in Individuals With Alcohol Dependence and Comorbid Anxiety or Depression
Brief Title: Acamprosate in Alcoholics With Comorbid Anxiety or Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Mclean Hospital (Other); Columbia University (Other)
Responsible Party: Principal Investigator, Susan Sonne, Associate Professor of Psychiatry, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CMP-MD-04
Record Dates: First submitted 2006-05-25; First posted 2006-05-26 (Estimated); Results first posted 2015-04-13 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-04

CONDITIONS: Alcohol Dependence; Major Depression; Social Anxiety Disorder; Generalized Anxiety Disorder
Keywords: Alcoholism; Mood; Anxiety; Acamprosate
MeSH Terms: conditions — Alcoholism; Depressive Disorder, Major; Phobia, Social; Generalized Anxiety Disorder; Anxiety Disorders | interventions — Acamprosate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Acamprosate tablets
  Interventions: Drug: Acamprosate
- 2 (Placebo Comparator): Matching placebo tablets
  Interventions: Drug: Acamprosate

INTERVENTIONS:
Drug: Acamprosate — 2 333mg tablets three times daily

SUMMARY:
STUDY OBJECTIVES:

The primary objective of this study is to compare the safety and efficacy of acamprosate versus placebo in the treatment of alcohol dependence in adults with co-occurring mood or anxiety disorders (specifically, depression (MDE), generalized anxiety disorder (GAD) or social anxiety disorder). Secondary objectives are to evaluate the effect of acamprosate treatment on mood and anxiety disorders.

STUDY DESIGN:

This is a randomized, double-blind, placebo-controlled trial evaluating acamprosate in the treatment of alcohol dependence in adult outpatients with concurrent mood and/or anxiety disorders. The active study phase will be 12 weeks in duration. There will be a two-week screening period, followed by 12 weeks of study medication and a follow-up assessment at 14 weeks from randomization.

STUDY POPULATION:

A total of 90 (30 per site) men and women aged 18-60 years who have a current diagnosis of alcohol dependence as well as a current DSM-IV diagnosis of either MDE, GAD and/or social anxiety will be recruited to participate in this study. Only those individuals whose psychiatric disorders are stable will be randomized to acamprosate or placebo. Three sites will participate in this trial.

TREATMENTS:

Eligible participants will be randomly assigned to receive either acamprosate or matching placebo for 12 weeks.

EFFICACY ASSESSEMENTS:

The primary efficacy outcome measure will be cumulative days abstinent as measured by self-report.

DETAILED DESCRIPTION:
Participants who meet all inclusion criteria and none of the exclusion criteria will be randomized to receive either acamprosate or placebo in a 1:1 ratio. Participants will be instructed to take (2) 333 mg tablets three times a day. Participants will be seen weekly for 12 weeks an again 14 weeks from randomization. At each weekly visit, participants will be asked about substance use and possible adverse events. They will also have their vital signs and weight measured at each visit. Psychiatric assessments, including the MADRS,HAM-A, Liebowitz Social Anxiety Scale, and Hospital Anxiety and Depression Scale will be performed at weeks 2, 4, 8, and 12. Alcohol craving will be assessed using the Obsessive Compulsive Drinking Scale at baseline and monthly. A urine drug screen will also be performed monthly. A clinical global impressions scale will be completed for both psychiatric and alcohol abuse symptoms at every visit. A breath alcohol test will be performed at every visit, and a urine drug screen will be performed at baseline and monthly during the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ages 18-60
2. Meet DSM-IV criteria for current (past 90 days) alcohol dependence
3. Must identify alcohol as the primary substance of abuse
4. Meet DSM-IV criteria for a current major depressive episode, GAD and/or social anxiety disorder
5. Have a stable psychiatric condition, as evidenced by a baseline CGI change score of 4 or below between the time of initial screening and the baseline visit, and if receiving psychotropic medication, must have a stable dose of medication for at least one month prior to baseline.
6. Must have a negative urine drug screen at the baseline visit; UDS may be repeated no more that twice to obtain an negative UDS
7. May be receiving medication treatment for anxiety/mood disorder as long as the dosage has been stable for 4 weeks prior to randomization.
8. May be engaged in psychosocial treatment for alcohol dependence or for mood/anxiety disorders.
9. Must abstain from alcohol for at least 3 consecutive days but no more than 21 days prior to medication initiation
10. Subjects must be able to adequately provide informed consent and function at an intellectual level sufficient to allow the accurate completion of all assessment instruments
11. Subjects must consent to random assignment, be willing to commit to medication treatment and follow-up assessments
12. CIWA-Ar scale is 8 or less at the baseline visit

Exclusion Criteria:

1. Individuals with a primary psychotic disorder or bipolar disorder
2. Individuals who meet DSM-IV criteria for current (past 90 days) dependence on substances other than alcohol, caffeine or nicotine
3. Individuals with an uncontrolled neurologic condition that could confound the results of the study
4. Individuals with an uncontrolled medical condition that may adversely affect the conduct of this trial or jeopardize the subject's safety
5. Regular use of benzodiazepines for the treatment of psychiatric symptoms (as defined as more than 12 times in the month prior to the screening visit)
6. Individuals receiving pharmacotherapy (e.g. disulfiram or naltrexone) for prevention of alcohol relapse
7. Women of childbearing potential who are lactating or refuse to use adequate forms of birth control
8. Current suicidal or homicidal risk

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2006-04; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan C Sonne, PharmD, BCPP, Principal Investigator — Medical University of South Carolina; Jennifer S Potter, PhD, Principal Investigator — Mclean Hospital; Richard Rosenthal, MD, Principal Investigator — Columbia University College of Physicians & Surgeons
Locations (3):
- United States (3):
  - McLean Hospital, Belmont, Massachusetts
  - Columbia University College of Physicians & Surgeons, New York, New York
  - Behavioral Health Services of Pickens County, Pickens, South Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from May 2006 to June 2008. The study was conducted at three sites including a rural community treatment program in South Carolina, an urban community treatment program in New York City, and at an academic setting at McLean Hospital in Belmont, MA
Groups:
- Acamprosate: Acamprosate tablets
- Placebo: Matching placebo tablets
Period: Overall Study
Arm/Group | Acamprosate | Placebo
Started | 45 | 45
Completed | 23 | 26
Not Completed | 22 | 19
Not completed — Withdrawal by Subject | 7 | 7
Not completed — Lost to Follow-up | 4 | 1
Not completed — Clinical deterioration | 1 | 2
Not completed — Excessive missed visits | 3 | 8
Not completed — Miscellaneous reasons | 7 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acamprosate | Placebo | Total
Number analyzed (Participants) | 45 | 45 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 45 | 45 | 90
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.6 (9.9) | 44.6 (8.7) | 44.1 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 19 | 35
  Male | 29 | 26 | 55
Region of Enrollment [Number; unit: participants]
  United States | 45 | 45 | 90

OUTCOME MEASURES:

1. Primary Outcome: Percent Days Drinking
Description: Drinking was assessed using the timeline followback (TLFB), which is a calendar-based instrument used to assess drinking and other substance use on a daily basis.
Time Frame: 12 weeks
Population: The primary outcome measure is difference in cumulative days abstinent. Based on the meta-analysis by Mann et al (2004). A total sample of 90 participants would be able to detect a difference of 11 (+/- 18) days between acamprosate and placebo groups with 80% power, and Type 1 error rate of 0.05.
Measure: Mean (Standard Error); unit: percentage of days drinking
Arm/Group | Acamprosate | Placebo
Number analyzed (Participants) | 45 | 45
percentage of days drinking | 34.9 (0.04) | 31.9 (0.04)
Statistical Analysis 1: Comparison: Acamprosate vs Placebo; Drinking outcomes were analyzed using multiple linear regression, controlling for site and baseline drinking level. Drinking and psychiatric symptoms assessed over time were examined using repeated measures (intercept only) mixed linear models (PROC MIXED in SAS). Analyses were performed using SAS statistical software (version 9.2; SAS Institute, Inc., Cary, NC). All tests were two-tailed and p-values less than 0.05 were considered statistically significant; Test type: Superiority or Other; p = 0.64, Mixed Models Analysis

2. Secondary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS)
Description: This 10-item rating scale is commonly used in the European pharmacotherapy trials, and it may have benefit in assessing substance abusers, because it focuses on cognitive symptoms of depression instead of the physical symptoms, which could be due to substance use and withdrawal (Yonkers and Samson, 2000). Total scores are used; Scale range is 0-60, with higher scores reflecting more severe symptoms.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Acamprosate | Placebo
Number analyzed (Participants) | 45 | 45
units on a scale | 11.0 (0.79) | 11.5 (0.76)

3. Secondary Outcome: Liebowitz Social Anxiety Scale
Description: The LSAS is a 24-item semi-structured clinician-administered instrument that assesses social anxiety through the evaluation of fear and avoidance of different social and performance situations. There are two subscales (avoidance and fear), with scores ranging from 0-72; Total score for instrument ranges from 0-144. This study only reports on total score. Higher scores reflect greater anxiety symptoms.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Acamprosate | Placebo
Number analyzed (Participants) | 45 | 45
units on a scale | 22.5 (3.09) | 23.2 (30.5)

4. Secondary Outcome: Hospital Anxiety and Depression Scale
Description: This is a 14-item self report assessment that contains two subscales (depression and anxiety) with each subscale ranging from 0-21; the total score ranges from 0-42. We report total scores. Higher scores represent worse symptoms.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Acamprosate | Placebo
Number analyzed (Participants) | 45 | 45
units on a scale | 10.5 (0.87) | 9.4 (0.84)

ADVERSE EVENTS:
Arm/Group | Acamprosate | Placebo
Serious Adverse Events (participants affected / at risk) | 1/45 | 1/45
Other Adverse Events (participants affected / at risk) | 25/45 | 21/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acamprosate (N=45) | Placebo (N=45)
Clinical Deterioration (Psychiatric disorders) | 1 (1) | 1 (1) — One participant in the placebo group experienced suicidal ideation and was hospitalized; one participant in the acamprosate group had worsening of alcohol use and was put in a higher level of care
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Acamprosate (N=45) | Placebo (N=45)
Headache (General disorders) | 13 (15) | 16/37 (20)
Diarrhea (Gastrointestinal disorders) | 7 (7) | 10 (10)
Nausea (Gastrointestinal disorders) | 5 (5) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No